CLINICAL TRIAL: NCT05795712
Title: 'Real Life' Monitoring of COPD Patients According to the 2017 GOLD Recommendations: Role of Bronchial Inflammation in Patient Management.
Brief Title: 'Real Life' Monitoring of COPD no ICS Patients
Acronym: COPDnoICS
Status: Completed | Type: Observational
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Responsible Party: Principal Investigator, RicercaTradate, Professor Antonio Spanevello, Istituti Clinici Scientifici Maugeri SpA
Other Study IDs: 2126 CE
Record Dates: First submitted 2023-03-09; First posted 2023-04-03 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — induced sputum blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Therapy Change from Baseline — The patient will be followed up from the point of view of therapy according to symptoms and flare-ups irrespective of systemic or peripheral eosinophil assessment

SUMMARY:
The aim of the study will be to assess in patients with mild-to-moderate COPD the role of inflammation in the patient's therapeutic management and follow-up.

DETAILED DESCRIPTION:
Studies have already shown that the risk of severe exacerbations in patients with COPD is associated with eosinophilic inflammation (1) and that patients with this type of inflammation have an increased risk of exacerbations if ICS administration is discontinued (2), but this indication does not appear in the latest GOLD recommendations to date.

The aim of the study will be to evaluate in patients with mild-to-moderate COPD the role of induced sputum and peripheral inflammation in the patient's therapeutic management and follow-up. For this purpose, the investigators will assess inflammation at the bronchial and systemic level by induced sputum and haemochrome at time 0 (recruitment), after 6,12, 18 and 24 months after therapy administration according to the updated 2017 GOLD recommendations.

ELIGIBILITY:
Inclusion Criteria:

* COPD diagnosis according to GOLD 2017 recommendations in clinical stability phase
* Post bronchodilator FEV1 ≥50 and ≤80
* Both smoker and ex-smoker
* Patients on LABA or LABA/LAMA therapy
* Patients also on ICS therapy discontinued at least 30 days after enrolment
* Patient able to cooperate with the required procedures
* Patient who has signed the informed consent

Exclusion Criteria:

* - Acute respiratory episode treated with antibiotics and/or steroids in the lower 4 weeks prior to enrolment
* Patients on roflumilast therapy
* Any exacerbation of COPD within 1 month after visit 1. A patient must not have had any hospitalisation for COPD within 6 months prior to visit 1.
* Comorbidities. History or current evidence of a clinically significant comorbidity or history of a positive test for HIV, hepatitis B or hepatitis C.
* History of adverse reactions including immediate or delayed hypersensitivity to any beta2-agonists,
* sympathomimetic drugs or any intranasal, inhaled or systemic corticosteroid therapy known or suspected sensitivity to the components of the inhalers used in the study (e.g. lactose in dry powder inhalers).
* Use of immunosuppressive drugs within 12 weeks prior to visit 1 and during the study, including use of systemic corticosteroids.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with COPD diagnosis in therapy with LABA or LAMA or LABA/LAMA
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2017-06-28 (Actual); Primary Completion 2020-09-07 (Actual); Study Completion 2023-03-09 (Actual)

PRIMARY OUTCOMES:
Number of participants which introduced ICS therapy after 24 month of follow up | 24 months
  The aim of our study will be to evaluate in patients with mild-to-moderate COPD the role of inflammation in the patient's therapeutic management and follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Istituti Clinici Maugeri Pneumologia, Tradate, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: Undecided